CLINICAL TRIAL: NCT03435003
Title: Designing Optimal Prevention and Management of Postoperative Nausea and Emesis for Patients Undergoing Laparoscopic Sleeve Gastrectomy
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Stony Brook University (Other)
Responsible Party: Principal Investigator, Konstantinos Spaniolas, Associate Professor of Surgery, School of Medicine Bariatric, Foregut and Advanced GI Surgery, Stony Brook University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 1074296-3
Record Dates: First submitted 2017-08-14; First posted 2018-02-15 (Actual); Results first posted 2024-02-14 (Actual); Last update posted 2024-02-14 (Actual); Status verified 2024-02

CONDITIONS: Post-operative Nausea and Vomiting; Laparoscopic Sleeve Gastrectomy
Keywords: Bariatric Procedure
MeSH Terms: conditions — Vomiting | interventions — Aprepitant; Scopolamine; Dexamethasone; Ondansetron; Metoclopramide; Prochlorperazine; Sugammadex; Propofol; Dexmedetomidine; Fentanyl; Sevoflurane; Desflurane

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention Arm (Experimental): A) Pre-operatively: aprepitant 80 mg oral capsule and scopolamine transdermal patch.
  B) Intra-operatively: total intravenous anesthesia (TIVA) will be maintained with IV infusions of propofol, and dexmedetomidine infusion or intermittent bolus dosing of fentanyl after induction. Sugammadex (2-4 mg/Kg IV) will be used for reversal of neuromuscular blockade in both groups. A single dose of dexamethasone 8 mg IV will be administered after induction, and a single dose of ondansetron 4 mg IV will be administered approximately 20 minutes prior to the end of operation.
  C) Post-operatively: Scheduled ondansetron and Raglan every 6 hours, using Compazine as a rescue medication.
  Interventions: Drug: Aprepitant 80 mg Oral Capsule; Drug: scopolamine transdermal; Procedure: Total intravenous anesthesia; Drug: Dexamethasone; Drug: Ondansetron; Drug: Reglan; Drug: Compazine; Drug: Sugammadex; Drug: Propofol; Drug: dexmedetomidine; Drug: Fentanyl
- Control Arm (Active Comparator): A) Pre-operatively: No intervention
  B) Intra-operatively: inhalation anesthetics (sevoflurane or desflurane) and intermittent opioid boluses will be used for maintenance of anesthesia, as standard practice in the institution of the investigators and across the country. PONV prevention measures in the control group will be limited to dexamethasone 8 mg and ondansetron 4 mg.
  C) Post-operatively: Scheduled ondansetron and Raglan every 6 hours, using Compazine as a rescue medication.
  Interventions: Drug: Dexamethasone; Drug: Ondansetron; Drug: Reglan; Drug: Compazine; Drug: Sugammadex; Drug: Sevoflurane; Drug: Desflurane

INTERVENTIONS:
Drug: Aprepitant 80 mg Oral Capsule — aprepitant 80 mg orally one hour prior to scheduled surgery
  Other Names: Emend
  Arms: Intervention Arm
Drug: scopolamine transdermal — scopolamine transdermal patch one hour prior to scheduled surgery
  Other Names: Transderm Scop
  Arms: Intervention Arm
Procedure: Total intravenous anesthesia — Maintenance of anesthesia without the use of inhaled anesthetics.
  Arms: Intervention Arm
Drug: Dexamethasone — Dexamethasone 8 mg intraoperatively
Drug: Ondansetron — Ondansetron 4 mg intraoperatively. Ondansetron will be given twice. Once intraoperatively and then post- operatively.
  Other Names: Zofran
Drug: Reglan — Postoperatively scheduled Reglan
  Other Names: Metoclopramide
Drug: Ondansetron — Postoperatively scheduled ondansetron
  Other Names: Zofran
Drug: Compazine — Postoperatively as needed compazine for breakthrough PONV
  Other Names: Compro
Drug: Sugammadex — Reversal with sugammadex
  Other Names: Bridion
Drug: Propofol — Intravenous anesthesia will be maintained through IV propofol
  Other Names: Diprivan
  Arms: Intervention Arm
Drug: dexmedetomidine — maintenance of anesthesia in the intervention arm
  Other Names: Precedex
  Arms: Intervention Arm
Drug: Fentanyl — intermittent bolus dosing of fentanyl will be used after induction for anesthesia maintenance
  Arms: Intervention Arm
Drug: Sevoflurane — inhalational anesthesia
  Other Names: Ultane
  Arms: Control Arm
Drug: Desflurane — inhalational anesthesia
  Arms: Control Arm

SUMMARY:
Bariatric surgery remains the most effective therapy for obesity. Postoperative nausea and vomiting (PONV) are commonly reported following bariatric surgery. The proposed study focuses on the most common bariatric procedure performed, laparoscopic sleeve gastrectomy (LSG), and aims to assess the effect of a post-operative nausea and vomiting-specific intervention. The investigators hypothesize that the intervention group will experience a reduction of nausea-related prolonged hospital stay and significantly improve patient-reported quality of recovery from surgery and quality of life.

DETAILED DESCRIPTION:
To test this hypothesis, participants undergoing sleeve gastrectomy will be randomized to two groups: control vs Nausea specific-intervention group. All subjects will be assessed with a nausea specific questionnaire at 1, 4, 12, 24 hours and 3 weeks after surgery. Patient satisfaction with recovery will be assessed using specialized questionnaires at baseline, 24 hrs. and 3 weeks following surgery. Serial assessments of nausea, vomiting, quality of life and quality of recovery, will allow the investigators to identify an effect on incidence and severity of Post-operative Nausea and Vomiting. Importantly, the investigators will evaluate for an impact in patient-reported measures of quality of life.

The total sample size is 83. This study will provide valuable insight on the epidemiology of post-operative nausea and vomiting after hospital discharge following Sleeve gastrectomy, which is currently poorly characterized. By allowing the investigators to assess the overall incidence of nausea and vomiting at different time points, this study will afford the opportunity to identify a time period of high incidence and further adjust our prevention efforts accordingly in future studies.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (18 years and older) undergoing LSG

Exclusion Criteria:

* Allergy to medications delineated in the protocol (muscle blockade, anesthetics, reversal agents)
* Inability to provide informed consent
* History of chronic nausea and emesis requiring medication
* Poorly controlled diabetes (HgA1c>9 mg/dl),
* History of previous bariatric or gastro-esophageal surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 83 (Actual)
Dates: Start 2017-08-28 (Actual); Primary Completion 2019-03-30 (Actual); Study Completion 2019-04-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Konstantinos Spaniolas, MD, Principal Investigator — Stony Brook University
Locations (1):
- Stony Brook University Hospital, Stony Brook, New York, United States

REFERENCES:
- [Derived] Naeem Z, Nie L, Drakos P, Yang J, Gan TJ, Pryor AD, Spaniolas K. The Relationship Between Postoperative Nausea and Vomiting and Early Self-Rated Quality of Life Following Laparoscopic Sleeve Gastrectomy. J Gastrointest Surg. 2021 Aug;25(8):2107-2109. doi: 10.1007/s11605-021-04923-4. Epub 2021 Feb 2. No abstract available. PMID 33528788

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Intervention Arm | Control Arm
Started | 41 | 42
Completed | 41 | 42
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Intervention Arm | Control Arm | Total
Number analyzed (Participants) | 41 | 42 | 83
Age, Continuous [Mean (Standard Deviation); unit: years] | 41.3 (9.7) | 43 (13) | 42.2 (11.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 26 | 29 | 55
  Male | 15 | 13 | 28
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 29 | 33 | 62
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 12 | 9 | 21
Previous history of postoperative nausea and vomiting (PONV) [Count of Participants; unit: Participants] | 0 | 0 | 0
Weight [Mean (Standard Deviation); unit: lbs] | 292 (52) | 293 (61) | 292.5 (56.4)
BMI [Mean (Standard Deviation); unit: kg/m2] | 47.3 (6.4) | 46.4 (7.5) | 46.8 (6.9)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With PONV-related Delay of Hospital Discharge
Description: The primary outcome would be incidence of PONV-related delay of hospital discharge following laparoscopic gastrectomy. Based on the current clinical pathway, patients are expected to be discharged on postoperative day 1 (day after surgery). A delay in discharge due to PONV will be the primary outcome.
Time Frame: up to 1 week post-operation (up to 2 weeks from baseline)
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention Arm | Control Arm
Number analyzed (Participants) | 41 | 42
Participants | 0 | 4

2. Secondary Outcome: Severity of PONV Measured Using a 10-point Verbal Rating Scale.
Description: The severity of PONV will be measured using a visual analogue scale. [0-10] The higher the value, the worse the outcome.
Time Frame: Baseline, 1 hour, 4 hours, 12 hours, 24 hours and 3 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention Arm | Control Arm
Number analyzed (Participants) | 39 | 40
score on a scale
  Baseline | 0.12 (0.56) | 0.10 (0.43)
  1 hr | 2.29 (2.86) | 3.68 (3.45)
  4 hr | 1.46 (1.82) | 2.76 (2.97)
  12 hr | 0.69 (1.47) | 2.19 (2.63)
  24 hr | 0.44 (1.16) | 1.80 (2.89)
  3 week | 0.15 (0.43) | 0.58 (1.68)

3. Secondary Outcome: Severity of PONV Measured Using the Rhodes Index
Description: The Rhodes Index of Nausea, Vomiting, and Retching (R-INVR) is a validated instrument used to measure the severity of Post-Operative Nausea and Vomiting (PONV). The index comprises eight items, each scored on a scale of 0 to 4, allowing for a total score range of 0 to 32 points .
  The scoring of each item on the Rhodes Index is as follows:
  0 points represent a minimum level of disturbance, 4 points represent a maximum level of disturbance . The total score from these eight items is summed to represent the severity of PONV, with higher scores indicating worse PONV experience. The index encompasses three subscales named "experience," "occurrence," and "distress" . Each of these subscales contributes to the total score to provide a comprehensive measure of PONV severity. Any score above zero on the R-INVR indicates that the participant experienced nausea .
Time Frame: Baseline, 1 hour, 4 hours, 12 hours, 24 hours and 3 weeks
Measure: Mean (Full Range); unit: score on a scale
Arm/Group | Intervention Arm | Control Arm
Number analyzed (Participants) | 40 | 42
score on a scale
  Baseline | 0.08 [0 to 3] | 0.19 [0 to 4]
  12 hr | 1.79 [0 to 8] | 6.17 [0 to 24]
  24 hr | 0.69 [0 to 6] | 5.26 [0 to 23]
  3 weeks | 0.13 [0 to 3] | 1.42 [0 to 4]

4. Secondary Outcome: Quality of Recovery Measured Using the Quality of Recovery QoR-15 Survey
Description: The quality of recovery-15 (QoR-15) is a patient-reported outcome measurement measuring QoR after surgery and anesthesia. The scale is arbitrary and ranges from 0 to 150. The higher the score, the worse the outcome.
Time Frame: 24 hours and 3 weeks
Measure: Mean (Full Range); unit: score on a scale
Arm/Group | Intervention Arm | Control Arm
Number analyzed (Participants) | 40 | 42
score on a scale
  24 hr | 120.59 [86 to 147] | 109.29 [59 to 146]
  3 weeks | 137.53 [78 to 150] | 130.64 [61 to 150]

5. Secondary Outcome: GI Specific Quality of Life Using the Gastrointestinal Quality of Life (GIQLI) Survey
Description: The GIQLI is a 36-item patient reported outcomes instrument designed to assess GI-specific health-related quality of life in clinical practice and clinical trials of patients with GI disorders. It has five domains (GI symptoms, emotion, physical function, social function and medical treatment) and sub-scores range from 0-4 while the total score range from 0-144. Higher scores mean better GI health-related quality of life.
Time Frame: Baseline, 24 hours and 3 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention Arm | Control Arm
Number analyzed (Participants) | 41 | 42
score on a scale
  Baseline | 108.34 (12.49) | 107.52 (13.35)
  3 Weeks | 100.71 (20.60) | 98.03 (25.22)

6. Secondary Outcome: Overall Quality of Life Using the EuroQol- 5 Dimension (EQ-5D) Instrument
Description: EQ-5D Descriptive System:
  Dimensions: Includes five dimensions: mobility, self-care, usual activities, pain/discomfort, anxiety/depression.
  Levels: Each dimension has 5 severity levels:
  1. No problems
  2. Slight problems
  3. Moderate problems
  4. Severe problems
  5. Extreme problems
  Time Frame: Assessed at baseline, 24 hours post-baseline, and 3 weeks.
Time Frame: Baseline, 24 hours and 3 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention Arm | Control Arm
Number analyzed (Participants) | 41 | 42
Participants
  Baseline: Usual activities: None | 29 | 29
  Baseline: Usual activities: Slight | 7 | 8
  Baseline: Usual activities: Moderate | 3 | 5
  Baseline: Usual activities: Severe | 2 | 0
  Baseline: Usual activities: Unable | 0 | 0
  Baseline: Usual activities: Not Reported | 0 | 0
  Baseline: Anxiety/depression: None | 26 | 29
  Baseline: Anxiety/depression: Slight | 11 | 10
  Baseline: Anxiety/depression: Moderate | 4 | 2
  Baseline: Anxiety/depression: Severe | 0 | 1
  Baseline: Anxiety/depression: Unable | 0 | 0
  Baseline: Anxiety/depression: Not Reported | 0 | 0
  Baseline: Mobility: None | 36 | 29
  Baseline: Mobility: Slight | 2 | 6
  Baseline: Mobility: Moderate | 2 | 6
  Baseline: Mobility: Severe | 1 | 1
  Baseline: Mobility: Unable | 0 | 0
  Baseline: Mobility: Not Reported | 0 | 0
  Baseline: Pain/discomfort: None | 24 | 20
  Baseline: Pain/discomfort: Slight | 12 | 13
  Baseline: Pain/discomfort: Moderate | 4 | 6
  Baseline: Pain/discomfort: Severe | 0 | 3
  Baseline: Pain/discomfort: Unable | 1 | 0
  Baseline: Pain/discomfort: Not Reported | 0 | 0
  Baseline: Self-care: None | 37 | 38
  Baseline: Self-care: Slight | 2 | 3
  Baseline: Self-care: Moderate | 1 | 1
  Baseline: Self-care: Severe | 1 | 0
  Baseline: Self-care: Unable | 0 | 0
  Baseline: Self-care: Not Reported | 0 | 0
  24 h: Usual activities: None | 11 | 15
  24 h: Usual activities: Slight | 13 | 9
  24 h: Usual activities: Moderate | 5 | 3
  24 h: Usual activities: Severe | 1 | 3
  24 h: Usual activities: Unable | 2 | 5
  24 h: Usual activities: Not Reported | 9 | 7
  24 h: Anxiety/depression: None | 29 | 25
  24 h: Anxiety/depression: Slight | 3 | 7
  24 h: Anxiety/depression: Moderate | 0 | 3
  24 h: Anxiety/depression: Severe | 0 | 0
  24 h: Anxiety/depression: Unable | 0 | 0
  24 h: Anxiety/depression: Not Reported | 9 | 7
  24 h: Mobility: None | 25 | 27
  24 h: Mobility: Slight | 6 | 3
  24 h: Mobility: Moderate | 1 | 3
  24 h: Mobility: Severe | 0 | 1
  24 h: Mobility: Unable | 0 | 1
  24 h: Mobility: Not Reported | 9 | 7
  24 h: Pain/discomfort: None | 4 | 4
  24 h: Pain/discomfort: Slight | 16 | 16
  24 h: Pain/discomfort: Moderate | 12 | 14
  24 h: Pain/discomfort: Severe | 0 | 1
  24 h: Pain/discomfort: Unable | 0 | 0
  24 h: Pain/discomfort: Not Reported | 9 | 7
  24 h: Self-care: None | 22 | 26
  24 h: Self-care: Slight | 5 | 4
  24 h: Self-care: Moderate | 4 | 3
  24 h: Self-care: Severe | 0 | 2
  24 h: Self-care: Unable | 1 | 0
  24 h: Self-care: Not Reported | 9 | 7
  3 weeks: Usual activities: None | 37 | 25
  3 weeks: Usual activities: Slight | 2 | 8
  3 weeks: Usual activities: Moderate | 0 | 3
  3 weeks: Usual activities: Severe | 1 | 0
  3 weeks: Usual activities: Unable | 0 | 0
  3 weeks: Usual activities: Not Reported | 1 | 6
  3 weeks: Anxiety/depression: None | 33 | 28
  3 weeks: Anxiety/depression: Slight | 6 | 6
  3 weeks: Anxiety/depression: Moderate | 1 | 1
  3 weeks: Anxiety/depression: Severe | 0 | 1
  3 weeks: Anxiety/depression: Unable | 0 | 0
  3 weeks: Anxiety/depression: Not Reported | 1 | 6
  3 weeks: Mobility: None | 37 | 27
  3 weeks: Mobility: Slight | 1 | 7
  3 weeks: Mobility: Moderate | 2 | 1
  3 weeks: Mobility: Severe | 0 | 1
  3 weeks: Mobility: Unable | 0 | 0
  3 weeks: Mobility: Not Reported | 1 | 6
  3 weeks: Pain/discomfort: None | 23 | 16
  3 weeks: Pain/discomfort: Slight | 14 | 13
  3 weeks: Pain/discomfort: Moderate | 2 | 6
  3 weeks: Pain/discomfort: Severe | 0 | 0
  3 weeks: Pain/discomfort: Unable | 1 | 0
  3 weeks: Pain/discomfort: Not Reported | 1 | 7
  3 weeks: Self-care: None | 38 | 31
  3 weeks: Self-care: Slight | 1 | 4
  3 weeks: Self-care: Moderate | 1 | 1
  3 weeks: Self-care: Severe | 0 | 0
  3 weeks: Self-care: Unable | 0 | 0
  3 weeks: Self-care: Not Reported | 1 | 6

ADVERSE EVENTS:
Time Frame: From enrollment until the participants 3 week follow up post-operative appointment.
Arm/Group | Intervention Arm | Control Arm
All-Cause Mortality (participants affected / at risk) | 0/41 | 0/42
Serious Adverse Events (participants affected / at risk) | 0/41 | 0/42
Other Adverse Events (participants affected / at risk) | 0/41 | 0/42

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2019-05-22): https://cdn.clinicaltrials.gov/large-docs/03/NCT03435003/Prot_SAP_002.pdf
  • Informed Consent Form (2018-05-10): https://cdn.clinicaltrials.gov/large-docs/03/NCT03435003/ICF_001.pdf